CLINICAL TRIAL: NCT00691639
Title: Collection of Blood Specimens From Patients in AL-3789 Studies for Elevated Intraocular Pressure (IOP)
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Alberta Davis, Alcon
Other Study IDs: C-07-27
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Open-Angle Glaucoma
Keywords: Open-angle glaucoma; IOP
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients who are or were participants in any Alcon AL-3789 study.
  Interventions: Other: Blood Collection Only

INTERVENTIONS:
Other: Blood Collection Only — Blood Collection Only

SUMMARY:
The objective of this study is to obtain blood samples from patients who are or were participants in any Alcon AL-3789 clinical trial. Association will be conducted to search for genetic markers in patients with glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be currently or previously enrolled in Alcon clinical study and received AL-3789

Exclusion Criteria:

* Age related

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received anecortave acetate treatment
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States